CLINICAL TRIAL: NCT00971971
Title: Assessment of a Protocol Aiming to Prevent Intradialytic Hypotension in Critically Ill Acute Kidney Injury Patients
Brief Title: Prevention of Intradialytic Hypotension in Acute Kidney Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Emerson Quintino de Lima MD, PhD, Associate Professor, Nephrology Division, São JOsé do Rio Preto Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10727-6
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-09

CONDITIONS: Acute Kidney Injury; Acute Renal Failure
Keywords: Hypotension; Acute renal failure; acute kidney injury; dialysis; ICU
MeSH Terms: conditions — Acute Kidney Injury; Hypotension | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Traditional SLED
  Interventions: Procedure: Standard SLED
- Profiling (Experimental): dialysate temperature reduction with Na and ultrafiltration (UF) profiling
  Interventions: Procedure: Dialysis

INTERVENTIONS:
Procedure: Dialysis — dialysate temperature (DT) reduction with Na and ultrafiltration (UF) profiling
  Arms: Profiling
Procedure: Standard SLED
  Arms: Control

SUMMARY:
Intradialytic hypotension (IH) is a major complication during acute hemodialysis. The aim of this study was to evaluate the effects of dialysate temperature (DT) reduction with Na and ultrafiltration (UF) profiling on hemodynamics of critically ill acute kidney injury (AKI) patients submitted to sustained low-efficiency dialysis (SLED).

ELIGIBILITY:
Inclusion Criteria:

* Acute renal failure with a need of dialysis.

Exclusion Criteria:

* Patients with basal serum creatinine > 3 mgdL.
* Patients submitted to renal transplantation.
* Patients unlikely to survive.
* Declination in authorization to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Intradialytic hypotension | At dialysis session

SECONDARY OUTCOMES:
Dialysis dose | dialysis session

CONTACTS AND LOCATIONS:
Locations (1):
- São Jose do Rio Preto Medical School, São José do Rio Preto, São Paulo, Brazil